CLINICAL TRIAL: NCT05243602
Title: Switching Virally Suppressed HIV-1 Infected Elderly Adults (Age ≥ 60 Years) Without Prior Confirmed Virological Failure From Current Anti-retroviral Regimen to Bictegravir, Emtricitabine and Tenofovir Alafenamide (B/F/TAF)
Brief Title: BFTAF Elderly Switch Study
Acronym: BFTAF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nairobi (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Loice Achieng, Principal Investigator, University of Nairobi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BFTAF
Record Dates: First submitted 2022-01-31; First posted 2022-02-17 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: HIV-1-infection
Keywords: HIV; Bictegravir; Tenofovir alafenamide; Switch; Elderly; Non-inferiority; First-line
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Intervention Model Description: Randomised, controlled open-label clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Switch to B/F/TAF (Experimental): Participants in this arm will switch from their current ARV regimen to the study drug B/F/TAF. This is an oral drug administered once daily for the duration of the study.
  Interventions: Drug: Switch to B/F/TAF
- Continue current regimen (Active Comparator): Participants in this arm will be maintained on their pre-enrollment ARV regimen for the duration of the study.
  Interventions: Drug: Continue current regimen

INTERVENTIONS:
Drug: Switch to B/F/TAF — This is a combined pill containing 50mg of bictegravir, 200mg of emtricitabine and 25mg of tenofovir alafenamide
  Other Names: Biktarvy
  Arms: Switch to B/F/TAF
Drug: Continue current regimen — Participants will continue taking the same ARV regimen they were on before enrollment with no change in drug or dosage for the duration of the trial
  Other Names: Control
  Arms: Continue current regimen

SUMMARY:
BACKGROUND: Current Kenya National Anti-retroviral (ARV) Guidelines and World Health Organization (WHO) Guidelines recommend first-line therapy of tenofovir disoproxil fumarate (TDF), lamivudine (3TC) and dolutegravir (DTG) for adult people living with HIV (PLHIV). This regimen has limitations, particularly for the aging PLHIV who are more likely to have pre-existing comorbidities and higher risk of developing comorbidities, including osteopenia, osteoporosis, and renal insufficiency. Abacavir, the preferred alternative nucleoside reverse transcriptase inhibitor (NRTI) in Kenya, is associated with increased cardiovascular risk that also limits its use in elderly populations. B/F/TAF is highly efficacious, well tolerated, co-formulated in a small pill, and does not have the same bone, renal or cardiovascular risks associated with currently recommended regimens in Kenya. We are not aware of any clinical trial to date that has been fully powered to compare ARV regimens for the increasing population of elderly PLHIV.

BROAD OBJECTIVE: We will compare the efficacy, safety, and impact on bone mineral density of switching to B/F/TAF to that of remaining on current ARV regimen in a population of elderly patients (60 years old or greater) with no prior confirmed treatment failure in Kenya.

DETAILED DESCRIPTION:
BACKGROUND

Kenya has the fourth largest burden of HIV globally with close to 1.5 million people living with HIV, with the highest prevalence seen in the age group 45-54 years. As PLHIV live longer with early and wider access to ART, we will have an increasingly aging population of PLHIV. The current Kenya National Guidelines and World Health Organization guidelines recommend TDF/3TC/DTG as the preferred first-line regimen for adults. This regimen is efficacious, available as a single-tablet regimen, is relatively well tolerated, and has a reasonable safety profile, particularly in younger populations.

Managing older populations is more challenging due to the presence of multiple comorbidities including cardiovascular disease, renal disease and bone disease. TDF is known to cause both renal insufficiency and osteoporosis/osteopenia, and is not recommended for patients with pre-existing renal disease or osteoporosis. Guidelines recommend measurement of renal function before initiation of TDF and ongoing monitoring of renal function, which is a potential barrier to rapid antiretroviral therapy (ART) initiation and is not always available or feasible in resource limited settings. Measurement of bone mineral density is expensive and not routinely carried out in resource-limited settings and osteoporosis is often only detected after a fracture. Elderly patients are more likely to have contraindications to the use of TDF but identifying those with contraindications is either not done or is costly and/or can result in a delay in treatment. The current alternative to TDF in many countries is abacavir (ABC), which is associated with an increased risk for cardiovascular events that is a particular concern for elderly patients, and has the disadvantage that it does not treat hepatitis B virus (HBV) co-infection.

RATIONALE

Tenofovir alafenamide (TAF) is a pro-drug of TDF whose pharmacokinetics allow for much lower dosing and reduced renal and bone toxicity compared to TDF, and is also approved to treat HBV. Switch from TDF to TAF has been associated with improvement in bone mineral density and reversion of osteoporosis.

Bictegravir is a highly efficacious integrase inhibitor that is non-inferior to DTG for naïve patients and those who are already virally suppressed on DTG/3TC/ABC. Clinical trials have also shown lower rates of drug-related adverse events with B/F/TAF compared to DTG/3TC/ABC or compared to a regimen comprising DTG, emtricitabine (FTC) and TAF (DTG+FTC/TAF). B/F/TAF is a single-tablet once-daily pill that is much smaller than other INSTI co-formulated pills, a fact that may be attractive to patients. The advantages of B/F/TAF are important for all PLHIV but particularly for the elderly population.

There is emerging data on increased weight gain associated with use of TAF, BIC or DTG, which may raise concerns about a potential increase in cardiovascular risk and development of type 2 diabetes for PLHIV treated with BFTAF.

TDF is known to have lipid-lowering effects and there is an association between increasing lipid parameters with a switch from TDF to TAF, without a difference in change in the total cholesterol to high-density lipoprotein (HDL) ratio.

A small retrospective cohort analysis found that switching virally suppressed PLHIV from TDF to TAF was associated with an increase in atherosclerotic cardiovascular disease (ASCVD) risk score, however there was no change in the total cholesterol to HDL ratio. A major limitation of this study was that it did not include a comparison group of non-switchers and it is not clear that the analysis adequately controlled for the known age-determined increase in ASCVD risk. Another retrospective cohort analysis of switching PLHIV from TDF to TAF similarly found an increase in lipid parameters without an increase in low-density lipoprotein to HDL ratio; ASCVD risk score was not analyzed. A post-hoc analysis of a prospective trial comparing PLHIV initiated on TDF vs TAF-containing regimens found a small but significantly greater increase in ASCVD risk scores in the TAF arm by week 96, however there was no difference in changes between risk categories.

In the ADVANCE trial, where ARV-naïve PLHIV were randomized to receive either TAF/FTC+DTG, TDF/FTC+DTG or a combination of TDF, FTC and efavirenz (EFV), there was a higher risk of cardiovascular disease (based on Framingham or QRISK scores) at week 48 with TAF/FTC+DTG compared to TDF/FTC/EFV, but no statistically significant difference in risk between TAF vs TDF within the DTG arms. This study also found that participants treated with TAF/FTC+DTG were at higher risk for developing type 2 diabetes than participants treated with TDF/FTC+DTG (based on QDiabetes risk scores).

We are not aware of any clinical trial to date that has been fully powered to compare ARV regimens for the increasing population of elderly PLHIV, nor of any study evaluating a potential change in lipid parameters, cardiovascular risk or risk of type 2 diabetes associated with regimen switch to BFTAF in an elderly population. We propose to conduct an open-label non-inferiority switch trial among elderly PLHIV to address this knowledge gap.

HYPOTHESES

1. Switch of virologically suppressed HIV-1 infected elderly adults (≥ 60 years) with no prior confirmed treatment failure to B/F/TAF is non-inferior to continuing current ARV regimen, as determined by risk of developing virological failure by 48 weeks
2. Switch to B/F/TAF will result in increased lumbar spine BMD relative to remaining on current ARV regimen among this elderly population

PRIMARY OBJECTIVES

1. To evaluate the non-inferiority of switching to B/F/TAF, compared to maintaining the current ARV regimen, in virologically suppressed HIV-1 positive elderly adults (≥ 60 years) with no prior confirmed virological failure, as determined by HIV-1 RNA polymerase chain reaction (PCR) ≥ 50 copies/ml at week 48
2. To evaluate the effect of B/F/TAF relative to maintaining the current ARV regimen on percentage change in lumbar spine bone mineral density (BMD) after 48 weeks as measured by dual-energy X-ray absorptiometry (DXA)

STUDY DESIGN

This is a phase IV, multi-center, two-arm, open-label, randomized trial over 48 weeks, describing the efficacy and safety of switching from current ARV regimen to B/F/TAF in virally suppressed HIV-1 infected elderly adults (≥ 60 years) who have been on ART for at least 24 weeks and having achieved virological suppression (HIV-1 RNA < 50 copies/ml) for at least 12 weeks, with no prior confirmed virological failure. Participants will be randomized at baseline to remain on their pre-enrollment ARV regimen or switch to B/F/TAF.

The study will take place at two sites in Kenya: Kenyatta National Hospital (KNH, the largest teaching and referral hospital in Kenya), and Jaramogi Oginga Odinga Teaching and Referral Hospital (JOOTRH, the largest teaching and referral hospital in the Nyanza region of Kenya). The outpatient HIV clinics at these sites currently provide ART to over 15,000 PLHIV combined, including over 1,000 elderly patients on first line ART (85% of whom are on TDF/3TC NRTI backbone combined with either DTG or EFV; no patients are currently on TAF or BIC).

Study visits will take place at screening, baseline, and weeks 4, 12, 24, 36, and 48 (with a 4-week extension as required for confirming HIV-1 RNA levels within the FDA snapshot window). HIV-1 RNA viral load will be performed at screening and weeks 4, 12, 24 and 48. If HIV-1 RNA is ≥ 50 copies/ml then a repeat test will be performed at least 2 weeks after the detectable result to confirm virological failure. If the repeat HIV-1 RNA result is ≥ 50 copies/ml this confirms protocol-defined virological failure (PDVF) and genotypic resistance testing will be performed for any repeat viral load ≥ 500 copies/ml. DXA of the lumbar spine and total hip will be performed at baseline and weeks 24 and 48 among the BMD monitoring population. Other routine study investigations will include cluster of differentiation 4 (CD4) count, complete blood count, serum creatinine (Cr), alanine aminotransferase (ALT), aspartate aminotransferase (AST), HBsAg, fasting lipids, fasting glucose and patient satisfaction questionnaires (HIVTSQ).

Participants will be randomized at baseline in a 1:1 ratio using a computer-generated randomization sequence to either continue with their current ARV regimen or switch to B/F/TAF.

STUDY POPULATION

Number of Participants and Participant Selection

The anticipated sample size is 516 participants (258 per study arm) started on study treatment among patients on ARV therapy for at least 24 weeks and no prior virological failure (defined as two consecutive HIV-1 RNA viral loads ≥ 50 copies/ml separated by at least 2 weeks), with a viral load of < 50 copies/ml for at least 12 weeks, and aged 60 years or above. Patients who have a prior history of changing ARV regimens for reasons other than treatment failure can participate in the study if they meet all eligibility criteria. We anticipate screening approximately 740 patients and enrolling 520 participants to achieve the sample size of 516 participants on treatment. There are currently over 1,000 elderly patients on first-line ARV therapy at the two study sites. Assuming a viral suppression rate of 85% among this group (MoH, 2019), we will have at least 850 patients available for screening in order to enrol the sample size 516 participants on treatment. The estimated enrollment per study site is: KNH, 330; JOOTRH, 190.

Participants enrolled at KNH will enter the BMD monitoring population (after excluding participants with pre-existing conditions likely to decrease validity of BMD estimates).

The primary analyses will use all participants in the intent-to-treat exposed (ITT-E) population, consisting of randomly assigned participants who receive at least one dose of the study drug.

Recruitment

Participants will be recruited from patients who are receiving routine outpatient HIV care at the two study sites. Eligible participants who provide written informed consent will undergo screening laboratory investigations (HIV-1 RNA viral load, complete blood count, AST, ALT, serum Cr, and HBsAg).

Patients who meet all eligibility criteria after screening investigations will be enrolled in the study within 28 days of the screening. During the enrollment visit, participants will be randomized in a 1:1 ratio to continue their current ARV regimen or switch to B/F/TAF.

Participants who enrol into the study at KNH will constitute the BMD monitoring population (after excluding participants with pre-existing conditions likely to decrease validity of BMD estimates), for whom baseline total hip and lumbar spine DXA will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to understand and comply with the protocol requirements, instructions and restrictions
* Able and willing to give informed consent
* Age 60 years or above
* Documented HIV-1 infection as confirmed by HIV-antibody testing as per the Kenya National Guidelines
* Has been receiving an ARV regimen for at least 24 weeks
* Documented HIV-1 RNA viral load < 50 copies/ml at least 12 weeks prior to enrollment and no viral rebound between the first viral load < 50 copies/ml and the screening viral load
* HIV-1 RNA viral load < 50 copies/ml at screening (within 28 days prior to enrollment)

Exclusion Criteria:

* Confirmed treatment failure as defined by two consecutive HIV-1 RNA viral loads ≥ 50 copies/ml separated by at least 2 weeks, after at least 6 months on ART or after a documented HIV-1 RNA viral load < 50 copies/ml
* Documented HIV-2 infection
* Using any concomitant therapy disallowed as per the reference safety information and product labeling for the study drugs
* Has AST and/or ALT at least 5-times greater than the upper limit of normal
* Has a creatinine clearance (CrCl) below 50 ml/min (as estimated using the Cockcroft-Gault estimate for glomerular filtration rate)
* Documented opportunistic infection within 4 weeks prior to the study enrolment
* Investigator opinion that the patient should switch or discontinue any ARV in their current regimen immediately for clinical reasons (e.g. anemia with Hb < 9.5 g/dl while currently on azathioprine (AZT); HBsAg positive without currently being on TDF or TAF plus 3TC or FTC; experiencing adverse events associated with any ARV in current regimen deemed significant enough to warrant immediate change in regimen)
* Any condition (including illicit drug use or alcohol abuse) or laboratory results which, in the investigator's opinion, interfere with assessments or completion of the study
* History or presence of allergy to the study drugs or their components
* BMD monitoring population will also exclude any participant with a pre-existing condition which is likely to decrease validity of bone mineral density estimations (including pre-existing vertebral or bilateral hip fractures, lytic or blastic metastases, bilateral hip arthroplasty, or lumbar spine internal fixation)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
Virologic failure at week 48 | 48 weeks
  Proportion of participants with HIV-1 RNA ≥ 50 copies/ml at week 48 (by US Food and Drug Administration (FDA) snapshot algorithm)
Change in BMD | 48 weeks
  Mean percentage change in lumbar spine BMD from baseline to week 48

SECONDARY OUTCOMES:
Virologic failure at week 24 | 24 and 96 weeks
  Proportion of participants with HIV-1 RNA ≥ 50 copies/ml at week 24
Treatment success | 24, 48 and 96 weeks
  Proportion of participants able to maintain virological suppression (HIV-1 RNA < 50 copies/ml with no discontinuation of the study treatment) at weeks 24 and 48
Change in BMD | 24 and 96 weeks
  Mean percentage change in lumbar spine BMD from baseline to week 24
Change in total hip BMD | 24, 48 and 96 weeks
  Mean percentage change in total hip BMD from baseline to weeks 24 and 48
Change in fracture risk as measured using the fracture risk assessment tool (FRAX) | 24, 48 and 96 weeks
  Fracture risk (FRAX) at weeks 24 and 48. Measure is a percentage with higher values indicating a greater risk of fracture
Change in patient satisfaction measured using the HIV treatment satisfaction questionnaire (HIVTSQ) | 24, 48 and 96 weeks
  Patient satisfaction scores at weeks 24 and 48 with scores ranging from 0 to 6, a higher score indicating greater satisfaction
Change in CD4 | 24, 48 and 96 weeks
  Change in CD4 count from baseline to weeks 24 and 48
Change in renal function | 24, 48 and 96 weeks
  Change in renal function (estimated glomerular filtration rate) from baseline to weeks 24 and 48
Change in total cholesterol | 24, 48 and 96 weeks
  Change in in total cholesterol at weeks 24 and 48
Change in low-density lipoprotein | 24, 48 and 96 weeks
  Change in low-density lipoprotein at weeks 24 and 48
Change in triglycerides | 24, 48 and 96 weeks
  Change in triglycerides at weeks 24 and 48
Change in total cholesterol to HDL ratio | 24, 48 and 96 weeks
  Change in total cholesterol to HDL ratio at weeks 24 and 48
Change in fasting blood glucose | 24, 48 and 96 weeks
  Change in fasting blood glucose at weeks 24 and 48
Laboratory and clinical adverse events | 24, 48 and 96 weeks
  Safety (laboratory and clinical adverse events) at weeks 24 and 48
Change in weight | 24, 48 and 96 weeks
  Change in weight from baseline to weeks 24 and 48
Change in body mass index | 24, 48 and 96 weeks
  Change in body mass index from baseline to weeks 24 and 48
Change in waist hip ratio | 24, 48 and 96 weeks
  Change in waist-hip ratio from baseline to weeks 24 and 48
Change in waist circumference | 24, 48 and 96 weeks
  Change in waist circumference from baseline to weeks 24 and 48
Type and frequency of genotypic resistance mutations | 24, 48 and 96 weeks
  List and frequency of genotypic resistance mutations for participants with protocol-defined virological failure and HIV-1 RNA PCR ≥ 500 copies/ml

CONTACTS AND LOCATIONS:
Overall Officials: Loice Achieng Ombajo, MD, MSc, Principal Investigator — University of Nairobi
Locations (2):
- Kenya (2):
  - Jaramogi Oginga Odinga Teaching and Referral Hospital, Kisumu
  - Kenyatta National Hospital, Nairobi

IPD SHARING:
Plan to Share IPD: Yes
We will share the individual patient data (IPD) that underlie the results reported after de-identification (text, tables, figures and appendices)
Supporting Information: Study Protocol
Time Frame: Beginning 6 months after publication of the final manuscript and for a period of 36 months
Access Criteria: Access to IPD will be subject to the University of Nairobi data sharing requirements. Written requests should be submitted to the Principal Investigator providing a brief description of the individual or group making the request and detailing the reason for the same. Prior to sharing the data, the requestor will be required to sign a data access and sharing agreement.